CLINICAL TRIAL: NCT02734992
Title: An Innovative Psychosocial Intervention for the Treatment of Chronic Pain Patients and Their Families
Brief Title: Acceptance and Commitment Therapy vs Medical Treatment as Usual Wait-list Control for Primary Headache Sufferers
Acronym: ALGEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cyprus (Other)
Collaborators: University of Crete (Other)
Responsible Party: Principal Investigator, Maria Karekla, Licensed Clinical Psychologist, Assistant Professor, Peer reviewed ACT trainer,, University of Cyprus
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: K3_K1_0
Record Dates: First submitted 2016-03-21; First posted 2016-04-12 (Estimated); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Headache
Keywords: Migraines; Tension-type Headache; Acceptance
MeSH Terms: conditions — Headache; Migraine Disorders; Tension-Type Headache

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acceptance and Commitment therapy + MTAU (Other): The Acceptance and Commitment therapy + MTAU (active treatment) consists of an unpublished manual developed for the purposes of the Algea project (Vasiliou & Karekla, 2015). The protocol specifies the following goals: (a) increase individuals' willingness to face uncomfortable internal experiences; b) promoting meaningful activities even in the present of head pain; (c) emphasizing acceptance as an alternative to avoidance in coping with headache; (d) clarifying individuals' values in important life domains; e) enhancing present moment-to-moment awareness.
  Participants will be asked to remain stable on their pharmacotherapy during this study. All eligible participants will be monitored (medication taken and amount) prior to the beginning of the intervention for three weeks to ensure stability of their conditions.
  Participants will complete questionnaires at pre-, post-treatment, and at 3-month follow-up. The WL group will enter treatment at the 3-month follow-up of the ACT-group.
  Interventions: Behavioral: ACT+ MTAU
- MTAU/ Wait-list Control Gr (Other): The MTAU/ Wait-list Control Gr will follow their usual treatments, including any new treatments their GPs or Neurologists might prescribe (mostly prophylactic and abortive medication), during the study at the time. Following the completion of the active group follow up 3months, participants allocated to the control group will receive the active treatment. Participants will complete the same questionnaires at three different time points: pre-, post-treatment, and at 3-month follow-up.
  Participants will be asked to remain stable on their pharmacotherapy during this study and inform the researchers of any changes. All eligible participants will be monitored (medication taken and amount) prior to the beginning of the intervention for three weeks to ensure stability of their conditions. Excluded participants will be referred to appropriate services.
  Interventions: Behavioral: Waitlist Control +MTAU

INTERVENTIONS:
Behavioral: ACT+ MTAU — Participants will be randomly assigned to one of the two groups: ACT-based intervention, plus their usual health care or Medical Treatment as Usual only (MTAU). The MTAU group will follow their usual medical treatment (prescribed headache medication). Treatment sessions will be conducted weekly by two co-therapists in groups of approximately 8-10 participants for 1 ½ hour. The control group will receive the ACT intervention following the completion of the 3-months follow-up assessment of the treatment group. Participants in both groups will complete primary and secondary outcome scales, as well as ACT process effects scales at pre, post and 3-months follow-up. The treatment group only will be also assessed at 6 and 12-months follow-up. The ACT protocol and the patients' workbook were developed for the needs of the Algea project (Vasiliou & Karekla, 2015). Techniques will focus on key ACT processes aiming at promoting psychological flexibility for the head pain experience.
  Other Names: The ALGEA STUDY
  Arms: Acceptance and Commitment therapy + MTAU
Behavioral: Waitlist Control +MTAU — Participants in the Waitlist control+ MTAU will not receive any active intervention. Upon completion of the 3 months follow-up assessment of the ACT+MTAU group, participants allocated in the Waitlist control+MTAU will receive the ACT intervention.
  Arms: MTAU/ Wait-list Control Gr

SUMMARY:
Research to date suggests that individuals with headache use avoidance as a way to manage their pain. Despite the wide use of avoidance as a coping mechanism of headache triggers, very little empirical evidence exist to support its effectiveness in headache management. New treatment approaches, such as Acceptance and Commitment Therapy (ACT), emphasize acceptance of headache and valued-living as alternatives to avoidance, have demonstrated preliminary support in helping individuals reduce headache-related disability and improve quality of life. Though, ACT has received empirical support for various chronic pain conditions, very little evidence exists as to its effectiveness for head pain problems. The current study will examine the efficacy of an ACT-based intervention, when added to medical treatment as usual (MTAU) vs. a waitlist control group across time (group differences at 3 months) and time changes for the ACT group at 12-months follow-up, on quality of life and general disability, among headache sufferers.

DETAILED DESCRIPTION:
The main behavioral treatment suggestion today for headache management is the prevention of headaches mostly via avoidance of external and internal headache triggers. Despite the wide use of avoidance in headache management, very little empirical evidence exists to support its effectiveness. Attempts at avoiding headache triggers or other internal private experiences associated with a headache, may increase trigger potency, restrict lifestyle, decrease internal locus of control, and exacerbate and maintain pain perception. New treatment approaches, such as Acceptance and Commitment Therapy (ACT), emphasize acceptance and valued living as alternatives to avoidance. Though ACT is an empirically supported treatment for chronic pain, there is limited evidence for its efficacy for head pain, and this evidence is afflicted with methodological limitations that need to be overcome before making conclusions as to the effectiveness of ACT for headaches. The purpose of the present study is to examine in a Randomized Controlled Trial (RCT) whether an ACT-based intervention for headache sufferers, added to Medical Treatment as Usual, decreases disability and improves the quality of life, compared to only Wait List Control (WL). Pre, post and 3-months group changes will be assessed. Patients participating in the ACT group will be monitored for a year period.

ELIGIBILITY:
Inclusion criteria:

1. meeting diagnostic criteria for Primary Headache based on the International Classification of Headache Disorders-II (beta version; 2013);
2. older than 18 years; c) sufficient Greek reading ability; and d) stable pharmacotherapy and headache experience (both remained unchanged for the past four weeks prior to assessment).

Exclusion criteria:

1. had an active psychotic spectrum condition or manic episode, suicidal ideation/intent or substance use problems (particularly misuse of prescription head pain relievers) within the past 6 months;
2. had a history of seizure, facial neuralgia or other secondary headache diagnoses (i.e., conditions that might preclude the accuracy of primary headache diagnosis);
3. scored <20 on the Mini-mental Status Examination suggesting significant cognitive impairment;
4. were living in nursing homes;
5. had multiple pain sides (pain experienced in multiple body sides or groups of muscles);
6. took part in other psychological interventions or counseling (particularly for managing headache) over the last two years;
7. were pregnant or lactating.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The Henry Ford Hospital Headache Disability Inventory (b-HDI; Jacobson, Ramadan, Aggarwal & Newman, 1994) | Group by time Changes from Baseline Headache Disability at 3 months follow-up
  b-HDI is a 25-item headache disability inventory assesses the effect of headaches on daily activities (e.g. 'Because of my headaches I am less likely to socialize') and emotional functioning (e.g. 'I feel desperate because of my headaches'). Items are divided into two sub-grouped scales: functional, representing the sensory component of headaches (e.g. intensity etc) (13-items); and emotional (12-items), representing the reactive or affective realm (Andrasik, Lipchik, McCrory, & Wittrock, 2005). The instrument is answered with "yes", "no" or "sometimes" and the higher the score the greater the disability caused by the headache. The b-HDI has shown high reliability (a=.84) and validity with other similar scales. For the purpose of this study, only the general headache disability score will be used, comprising of the two subscales.
The Migraine- Specific Quality of Life Questionnaire (MSQ v 2.1; Martin et al., 2000; under permission given by GlaxoSmithKline; GSK USMA health outcome group), | Group by time Changes from Baseline Headache Disability at 3 months follow-up
  The MSQ is a 14-items migraine-specific Likert-type scale assesses the impact of migraines on patients' quality of life over the past four weeks. The scale is divided into three dimensions: Role Restrictive (RR; 7 items), Role Preventive (RP; 4 items), and Emotional Function (EF; 3 items). Role- function restrictive describes the degree to which performance of daily activities are limited by migraines. Role Preventive (RP) assesses the amount of normal activities interrupted by migraines. The Emotional Function (EF) evaluates the degree of emotional effects of migraine (e.g., frustration, afraid and burden). Items ranged from 1 (none of the time) to 6 (all of the time). The revised MSQ (version 2.1) appears with sufficient psychometric validity and reliability (a coefficient= .86- .96), across different migraine groups (Cole, Lin & Rupnow, 2007; Rendas- Baum, Bloudek, Maglinte & Varon, 2013). For the purpose of this study the three dimensions will be used to assess functional changes.

SECONDARY OUTCOMES:
The Hospital Anxiety and Depression Scale (HADS; Zigmond, & Snaith, 1983) | Group by time Changes from Baseline Headache Disability at 3 months follow-up
  HADS is a 14 item questionnaire assessing levels of anxiety and depression symptomatology. Each subscale consists of 7 items rated on a 4-point scale (0-3). Higher scores indicate greater anxiety and depression. The Greek version presents with high internal consistency (Cronbach's alpha=.88) and validity (Michopoulos et al., 2008).
Greek Brief pain inventory: the pain severity subscale (G-BPI; Mystakidou, Mendoza, | Group by time Changes from Baseline Headache Disability at 3 months follow-up
  G-BPI is a 4-item scale rated in a Likert-type scale from 0= no pain to 10 = the most severe pain ever experienced. Ratings are taken for the present time and 24 hours prior to the interview. The G-BFI shows good internal consistency (a coefficient= .80) and sufficient validity. The Greek validity has also demonstrated a high reliability (a= .88 for severity) and sufficient validity with other similar instruments.
Number of visits to different physicians due to Headache (Adapted with permission from Vowles et al., 2008) | Group by time Changes from Baseline Headache Disability at 3 months follow-up
  articipants, will record the total number of HA-related medical visits had over the last two months at the time of the assessment (# HA- related visits to different physicians). Based on participant estimations, a summary score for number of different HA-related medical visits for HA will be calculated.
Number of medical utilization (# visits to primary care for HA, #visits to Emergency, #department for HA, # hospitalization due to HAs (adapted with permission from Vowles et al., 2008). | Group by time Changes from Baseline Headache Disability at 3 months follow-up
  Participants will record the total number of medical utilization had over the last two months at the time of the assessment, (# visits to primary care for HA, #visits to Emergency department for HA, # hospitalization due to HAs). Based on participant estimations, a summary score for number of medical utilization visits will be summed to provide an overall index of medical utilization related to HAs.

OTHER OUTCOMES:
The Chronic Pain Acceptance Questionnaire (G-CPAQ Greek adaptation; Vasiliou et al., 2017; Original McCracken et al, 2004) | Group by time Changes from Baseline Headache Disability at 3 months follow-up
  G-CPAQ is an 8 items measure, rated on a 7-point Likert scale (1=never true to 6=always true), assesses pain acceptance on two dimensions: (a) activity engagement: degree of engagement in meaningful activity even in the presence of pain and (b) pain willingness: degree of experiencing pain without trying to change, control, or struggle with it
Psychological inflexibility in pain scale (G-PIPS; Greek adaptation; Vasiliou et al., 2019; PIPS-II; Wicksell, Lekander, Sorjonen & Olsson, 2010) | Group by time Changes from Baseline Headache Disability at 3 months follow-up
  PIPS is a 12-item instrument of psychological inflexibility. PIPS-II contains two subscales: avoidance of pain (8 items) and cognitive defusion (4 items) related to pain. The avoidance subscale measures behaviors that lead to avoidance of pain, while the cognitive fusion subscale assesses how a patient's thoughts about an event can lead to avoidance of pain ( "I need to understand what is wrong in order to move on"). Responders rate answers on a 7-point Likert-type scale from "never true" (1) to "always true" (7). The scale has good psychometric properties, showing high reliability (a= .87) and sufficient construct validity as shown by relations with other constructs. Validation of the instrument in the Greek language shows similar with the original results (Vasiliou, Karekla, Michaelides, & Kasinopoulos, in preparation). The Greek version appears with high internal consistency (Cronbach's a= .80) and significant correlations with associated constructs.
Committed Action Questionnaire (CAQ; McCracken, Chilcot, & Norton, 2014), | Group by time Changes from Baseline Headache Disability at 3 months follow-up
  CAQ is an 8-item Likert-type scale assesses goals- directed behaviors (McCracken, 2014). It includes 13 positively worded items (e.g. "When a goal is difficult to reach, I am able to take small steps to reach it") and 11 negatively worded items (e.g. "I find it difficult to carry on with an activity unless I experience that it is successful") tapped into two related factors: positive and negative aspects of committed actions. Questions are ranged from 0 (never true) to 6 (always true) with higher scores denote higher committed actions. CAQ present with high internal consistency reliability (a= .87) and sufficient validity with other related instruments, including pain acceptance, depression, and functioning (McCracken et al., 2014).
The Valuing Questionnaire (VQ; Smoot et al.,2014) | Group by time Changes from Baseline Headache Disability at 3 months follow-up
  is a 10-item instrument, rated on a 7-point Likert scale (0=not at all true and 6=completely true), assessing the extent to which individuals act based on their personal values over the past week. The scale has two dimensions with 5 items each: progress in identified values (VQ-Pr) and obstruction of valued living (VQ-Ob). Higher scores in the progress subscale represent pursuing valued living, whereas higher scores on the obstruction subscale indicate the presence of psychological barriers (e.g., disturbing thoughts) in pursuing valued living.
The Cognitive Affective Mindfulness Scale-Revised (CAMS-R; Feldman et al., 2006) | Group by time Changes from Baseline Headache Disability at 3 months follow-up
  a 12-item questionnaire, rated on a 4-point Likert scale (1=rarely to 4=almost always), assessing affective and cognitive components of mindfulness. Higher scores reflect greater mindfulness levels or individual's ability to bring awareness on what is happening inside and around them, by fully engaging on the present moment with a non-judgmental way.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cyprus, Nicosia, Cyprus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vasiliou VS, Karademas EC, Christou Y, Papacostas S, Karekla M. Mechanisms of change in acceptance and commitment therapy for primary headaches. Eur J Pain. 2022 Jan;26(1):167-180. doi: 10.1002/ejp.1851. Epub 2021 Aug 18. PMID 34375444